CLINICAL TRIAL: NCT04621838
Title: To Evaluate the Safety and Performance of the AMS ActivHeal Silicone Foam and the ActivHeal Silicone Foam Lite Dressing With Respect to Wound Exudate Management, Wound Healing Progression and Peri Wound Skin Condition.
Brief Title: To Evaluate the Safety and Performance of the AMS ActivHeal Silicone Foam and the ActivHeal Silicone Foam Lite Dressing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: Cliniscience Sp. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WD2018-Silicone-02
Record Dates: First submitted 2020-10-09; First posted 2020-11-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-03

CONDITIONS: Wound
Keywords: Silicone Foams; Chronic wounds; Acute wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned intervention. (Experimental): Silicone Foam Dressing. Silicone Foam Lite.
  Subjects will undergo treatment of their chronic or acute wound as indicated in the instructions for use with Silicone Foam dressing and Silicone Foam Lite Dressing.
  Interventions: Other: Assigned interventions.

INTERVENTIONS:
Other: Assigned interventions. — Subjects will undergo treatment of their chronic and acute wounds as indicated in instructions for use, with Silicone Foam Dressing and Silicone Foam Lite Dressing.
  The patients will be evaluated at each dressing change over a six-week period (per Product) or until the wound is healed to extent that the use of the Silicone Foam and Silicone Foam Lite dressing is no longer indicated from the time that the patient has been recruited.

SUMMARY:
To demonstrate the safety and performance of both AMS ActivHeal Silicone Foam and AMS ActivHeal Silicone Foam Lite dressings to both the patient and clinician in managing both chronic and acute wounds.

DETAILED DESCRIPTION:
This PMCF study has been set up to investigate and assess residual risks in relation to the CE-marked AMS ActivHeal Silicone Foam and Silicone Foam Lite dressing . The purpose of this study is primarily to collect clinical follow-up data on the AMS ActivHeal Silicone Foam and Silicone Foam Lite dressing , as CE-marking was based on equivalence. The data and conclusions obtained from this study will be used to provide clinical evidence of safety and effectiveness for the clinical evaluation process.

ELIGIBILITY:
The patient population of this evaluation will consist of patients with either a chronic or acute wound of various wound types, according to the intended use of both the AMS ActivHeal Silicone Foam and ActivHeal Silicone foam lite dressing, and they meet study eligibility criteria.

Inclusion Criteria:

1. Males or females, age 18 years or above. (Females must not be pregnant and if of reproductive age should be using contraception).
2. Subjects who are able to understand and give informed consent to take part in the evaluation.
3. No local or systemic signs of infection, including new pain or increasing pain, erythema, local warmth, swelling, purulent discharge, pyrexia (in surgical wounds, typically five to seven days after surgery), delayed wound healing, abscess or malodour.
4. None to high levels of exudate

Exclusion Criteria:

1. Patients who decline the invitation to take part.
2. Patients who are known to be non-compliant with medical treatment,
3. Patients who are known to be sensitive to any of the dressing components.
4. Broken/ damaged or prone to blistering peri wound skin.
5. Presence of a clinically infected wound as determined by the presence of three or more of the following clinical signs: peri wound, erythema, pain between dressing changes, malodourous wound, abundant exudate, oedema, abscess, cellulitis, purulent discharge, discolouration, friable granulation tissue which bleeds easily.
6. Patients who have a current illness or condition which may interfere with wound healing in the last 30 days which may interfere with wound healing (carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse.)
7. Life expectancy of <6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Primary 1 Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to the management of wound exudate. | After each dressing change up to 6 weeks following application of dressing
  Success will be determined by no deterioration of the wound or peri wound skin. A relative score will be used to score maceration of zero (no maceration), one (minimal maceration), two (moderate maceration), and three (excessive maceration and need to withdraw patient from study.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to Wound Healing progression. | After each dressing change up to 6 weeks following application of dressing
  Success will be determined by no deterioration of the wound. The assessor will assess the wound size and the % tissue types within the wound.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to the per wound skin conditions. | After each dressing change up to 6 weeks following application of dressing
  Success will be determined by no deterioration of peri wound skin. The peri wound skin will be assessed for maceration and signs of inflammation. A relative score will be used to score maceration of zero (no maceration), one (minimal maceration), two (moderate maceration), and three (excessive maceration and need to withdraw patient from study). Success will be determined that over the evaluation an increased score would represent peri wound deterioration. This will be measured using VAS value (0= no erythema, redness and skin erosion and 10 = extensive erythema, redness and skin erosion).

SECONDARY OUTCOMES:
Effectiveness of dressing removal of both the Silicone Foam and Silicone Lite dressing will assessed. | After each dressing change up to 6 weeks following application of dressing
  The assessor will be required to record the pain score chosen by the patient pre removal of the dressing and record the pain score chosen by the patient during removal. Success will be determined by no increased in pain score and this will be measured using VAS value (0= no pain to 10= most pain imaginable).
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to wound pain. | After each dressing change up to 6 weeks following application of dressing
  Pain associated with the wound. The assessor will be required to record the pain score chosen by the patient and record the pain score chosen by the patient. Success will be determined by no increase in pain score and this will be measured using VAS value. (0= no pain to 10= most pain imaginable).
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to ease of use of the dressing. | After each dressing change up to 6 weeks following application of dressing
  Ease of use of the dressing. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to conformability of the dressing. | After each dressing change up to 6 weeks following application of dressing
  Conformability of the dressing. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to dressing contours to anatomical contours of major wound site. | After each dressing change up to 6 weeks following application of dressing
  Dressing contours to anatomical contours of major wound site. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to overall acceptability of the dressing. | After each dressing change up to 6 weeks following application of dressing
  Overall acceptability of the dressing. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to peri wound skin condition. | After each dressing change up to 6 weeks following application of dressing.
  Peri wound skin condition satisfaction. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to the management of exudate. | After each dressing change up to 6 weeks following application of dressing.
  Management of exudate satisfaction. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.
Effectiveness of both Silicone Foam and Silicone Lite dressing will assessed in regards to wound healing progression. | After each dressing change up to 6 weeks following application of dressing.
  Wound Healing Progression. The assessor will be required to rate their level of satisfaction. Success will be determined by no unsatisfied level of satisfaction, and this will be measured using the following 'highly satisfied', 'satisfied' or 'unsatisfied'.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Mikosiński, MD, PhD, Principal Investigator — Poradnia Chorób Naczyń Obwodowych MIKOMED; Katarzyna Rybołowicz, MD,PhD, Principal Investigator — Gabinet Ortopedyczny, Specjalistyczny Ośrodek Leczniczo-Badawczy,; Konrad Pańczak, MD,PhD, Principal Investigator — NZOZ Twój Lekarz Kobierzyce,
Locations (1):
- Poradnia Chorób Naczyń Obwodowych MIKOMED, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No